CLINICAL TRIAL: NCT05618912
Title: Scar Appearance After Postoperative Hydrocolloid Dressing Versus Standard Petrolatum Ointment: A Randomized Controlled Trial
Brief Title: Scar Appearance After Postoperative Hydrocolloid Dressing Versus Standard Petrolatum Ointment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Syril Keena Que, Assistant Professor of Clinical Dermatology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15768
Record Dates: First submitted 2022-10-23; First posted 2022-11-16 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Scar; Skin Scarring; Skin Cancer; Wound Heal; Wound of Skin; Surgical Wound; Patient Satisfaction; Patient Preference; Surgical Incision
Keywords: scar; dermatologic surgery; wound healing; wound of skin; skin cancer; surgical incision; patient satisfaction; patient preference; cosmetic outcome; scar appearance
MeSH Terms: conditions — Cicatrix; Skin Neoplasms; Surgical Wound; Patient Satisfaction; Patient Preference | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: Each patient will have the surgical scar treated with either type of intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- hydrocolloid dressing arm (Experimental): After informed consent and closing the wound with the sutures, the scar will be covered by a hydrocolloid dressing, which will be left in place for 7 days (Experimental)
  Interventions: Device: Hydrocolloid dressing
- Petrolatum jelly dressing arm (Active Comparator): and the other group of patients (control), after closing the wound with the sutures, the scar will be covered with petrolatum jelly during this time period, which has to be re-applied daily.
  Interventions: Other: Petrolatum jelly dressing

INTERVENTIONS:
Device: Hydrocolloid dressing — A single hydrocolloid dressing will be applied to the surgical site for 7 days following dermatologic surgery
  Arms: hydrocolloid dressing arm
Other: Petrolatum jelly dressing — The patient with the control wound will be covered with petrolatum jelly during this time period, which has to be re-applied daily.
  Arms: Petrolatum jelly dressing arm

SUMMARY:
Patients will be randomized either to receive standard daily dressing or hydrocolloid dressing using a randomization generator. After closing the wound with the sutures,the scar will be covered by a hydrocolloid dressing, which will be left in place for 7 days(Experimental) or the standard dressing (Control) that will be covered with petrolatum jelly and bandaging during this time period, which has to be re-applied daily. Patients and dermatologic surgeons will then complete surveys 7 days, 30 days, and 90 days after surgery to evaluate the cosmetic appearance of these scars.

ELIGIBILITY:
Inclusion Criteria:

1. Adult > 18 years of age
2. Linear scars
3. Patients underwent conventional excision or Mohs micrographic surgery for primary cutaneous cancer or other cutaneous condition that required surgical intervention

Exclusion Criteria:

1. Scar localization on acral or hair bearing sites
2. Patients unable to converse in English
3. Patients requiring flap or graft for closure of wound
4. History of allergy to adhesives
5. Patient using topical chemotherapy agents on the surgical site or planning to start it within 3 months after surgery
6. Use of hydrocolloid dressings for post-operative wound care in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Physicians Dermatology Meridian Crossing, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes SP, Rivera S, Hooper PB, Slaven JE, Que SKT. Hydrocolloid dressing versus conventional wound care after dermatologic surgery. JAAD Int. 2021 Dec 21;6:37-42. doi: 10.1016/j.jdin.2021.11.002. eCollection 2022 Mar. PMID 34993497
- [Derived] Bell MC, Gangodawila TW, Morr CS, Xue GR, Iqbal A, Merkel EA, Abdulhak AH, Slaven JE, Que SKT. Hydrocolloid Dressing vs Petroleum Ointment for Scar Appearance After Dermatologic Surgery: A Randomized Clinical Trial. JAMA Dermatol. 2025 Dec 1;161(12):1246-1251. doi: 10.1001/jamadermatol.2025.4051. PMID 41123900

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
Started | 72 | 74
Completed | 58 | 55
Not Completed | 14 | 19
Not completed — Lost to Follow-up | 14 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.5) | 61.3 (13.5) | 61.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 85
  Male | 32 | 29 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 72 | 73 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cosmetic Outcome
Description: Patient and surgeon assessment of cosmetic outcome using modified visual analogue scar scale. The minimum value is 1 and the maximum value is 10. 1 is the worst possible scar appearance and 10, is the best possible scar appearance.
Time Frame: 7 days
Population: The above numbers reflect the number of patients who responded at 7-day postoperative followup and is smaller than the original number of participants in each arm due to lack of response by some participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
Number analyzed (Participants) | 64 | 65
score on a scale
  Patients - Overall | 7.4 (2.0) | 6.6 (1.9)
  Surgeons - Overall | 6.3 (1.7) | 6.00 (1.8)
  Patients - Color | 7.1 (1.8) | 6.6 (1.8)
  Surgeons - Color | 6.44 (0.13) | 5.97 (0.14)
  Patients - Texture | 6.8 (2.0) | 6.4 (2.0)
  Surgeons - Texture | 5.83 (0.16) | 5.80 (0.15)
  Patients - Scar Line | 7.0 (2.1) | 6.4 (2.1)
  Surgeons - Scar Line | 6.48 (0.12) | 6.30 (0.12)

2. Primary Outcome: Cosmetic Outcome
Description: as for outcome 1
Time Frame: 30 days
Population: The above numbers reflect the number of patients who responded at 30-day postoperative followup and is smaller than the original number of participants in each arm and the number of participants analyzed at 7-day followup due to lack of response by some participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
Number analyzed (Participants) | 64 | 60
score on a scale
  Patients - Overall | 7.6 (1.5) | 7.6 (1.9)
  Surgeons - Overall | 7.07 (0.13) | 7.00 (0.14)
  Patients - Color | 7.5 (1.5) | 7.5 (1.8)
  Surgeons - Color | 7.17 (0.14) | 7.21 (0.15)
  Patients - Texture | 7.0 (1.6) | 6.4 (2.1)
  Surgeons - Texture | 6.48 (0.12) | 6.30 (0.12)
  Patients - Scar Line | 7.3 (1.7) | 7.3 (2.1)
  Surgeons - Scar Line | 7.04 (0.14) | 6.95 (0.14)

3. Primary Outcome: Cosmetic Outcome
Description: as for outcome 1
Time Frame: 90 days
Population: The above numbers reflect the number of patients who responded at 90-day postoperative followup and is smaller than the number of participants initially enrolled and the number analyzed at 7-day and 30-day followup due to lack of response by some participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
Number analyzed (Participants) | 58 | 55
score on a scale
  Patients - Overall | 8.2 (1.8) | 8.1 (1.6)
  Surgeons - Overall | 7.94 (0.12) | 7.92 (0.12)
  Patients - Color | 7.1 (1.8) | 6.6 (1.8)
  Surgeons - Color | 6.44 (0.13) | 5.97 (0.14)
  Patients - Texture | 8.1 (1.7) | 7.8 (2.0)
  Surgeons - Texture | 8.28 (0.11) | 8.14 (0.12)
  Patients - Scar Line | 8.1 (1.9) | 7.9 (2.1)
  Surgeons - Scar Line | 7.89 (0.13) | 7.86 (0.13)

4. Secondary Outcome: Number of Participants With Complications
Description: Complication rate including hematoma, seroma, wound infection requiring antibiotics, opening and drainage of wound, dehiscence. Complications will be assessed by physicians other than operating surgeon
Time Frame: 7 days, 30 days, 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
Number analyzed (Participants) | 72 | 74
Participants
  Itching | 29 | 28
  Surgical site pain | 14 | 7
  Required antibiotics | 0 | 0
  Wound dehiscence | 4 | 0
  Post-op bleeding | 13 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 90-day period following the patient's excisional surgery
Arm/Group | Hydrocolloid Dressing Arm | Petrolatum Jelly Dressing Arm
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/74
Other Adverse Events (participants affected / at risk) | 60/72 | 40/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocolloid Dressing Arm (N=72) | Petrolatum Jelly Dressing Arm (N=74)
Itching (Skin and subcutaneous tissue disorders) | 29 (29) | 28 (28) — Assessed via surveys sent to all patients in the trial
Surgical site pain (Skin and subcutaneous tissue disorders) | 14 (14) | 7 (7) — Assessed via surveys sent to all patients in the trial
Required antibiotics (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) — Assessed via surveys sent to all patients in the trial
Wound dehiscence (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — Assessed via surveys sent to all patients in the trial
Post-op bleeding (Skin and subcutaneous tissue disorders) | 13 (13) | 5 (5) — Assessed via surveys sent to all patients in the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT05618912/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT05618912/ICF_001.pdf